CLINICAL TRIAL: NCT07054905
Title: Prediction of Hyperkalemia in Dialysis Patients Through Waveform Analysis Using Wearable ECG
Status: Not yet recruiting | Type: Observational
Sponsor: Kyungho Park (Other)
Responsible Party: Sponsor-Investigator, Kyungho Park, Assistant Professor of Nephrology, Chungnam National University Hospital, Chungnam National University Hospital
Organization: Chungnam National University Hospital (Other)
Other Study IDs: CNUH 2025-05-023
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Hyperkalemia; Chronic Kidney Disease
Keywords: Wearable ECG; Hemodialysis; Potassium; HiCardi
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemodialysis Patients: Adults with chronic kidney disease receiving maintenance hemodialysis three times per week. Participants will wear a HiCardi single-lead wearable ECG device during dialysis sessions for 8 weeks. ECG data will be collected four times in coordination with routine blood potassium tests to evaluate the correlation between ECG waveform changes and hyperkalemia.
  Interventions: Device: HiCardi wearable ECG

INTERVENTIONS:
Device: HiCardi wearable ECG — A chest-attached, single-lead wearable ECG device used to collect real-time ECG data from hemodialysis patients. The device records ECG waveforms during dialysis sessions and transmits the data to a secure cloud platform. This non-invasive tool is used to analyze T-wave morphology for early detection of hyperkalemia in patients with chronic kidney disease.

SUMMARY:
This study aims to evaluate whether hyperkalemia, a potentially life-threatening condition in dialysis patients, can be detected early using a wearable single-lead ECG device. Patients with chronic kidney disease undergoing hemodialysis will wear a chest-attached ECG sensor (HiCardi) during dialysis sessions. ECG data will be collected four times over six weeks, in coordination with routine blood tests measuring serum potassium levels. The goal is to analyze changes in ECG waveforms, such as T waves, and determine if these correlate with elevated potassium levels. The study is non-interventional and observational, focusing on real-time, non-invasive monitoring. It is expected to improve clinical decision-making by enabling early detection of hyperkalemia without additional blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older
* Diagnosed with chronic kidney disease (CKD) and receiving maintenance hemodialysis three times per week
* Stable clinical condition without acute complications in the past 3 months
* Ability to understand and sign informed consent
* No physical or physiological barrier to wearing an ECG device

Exclusion Criteria:

* Significant skin conditions (e.g., severe dermatitis, burns) that prevent ECG device attachment
* Refusal or inability to comply with study procedures

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease undergoing regular hemodialysis at Chungnam National University Hospital. Participants are selected based on clinical stability and willingness to provide informed consent. The population includes both male and female adults without age restriction.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Correlation between EKG characteristics and serum potassium level | Week 0, Week 2, Week 4, Week 6
  The primary outcome is the correlation between EKG characteristics (e.g., T wave amplitude, QRS duration, P wave morphology) measured using a wearable single-lead ECG device and serum potassium levels obtained from blood tests. Data will be collected at four time points over 8 weeks.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the data include sensitive clinical and biometric information that may risk participant privacy. In addition, there is no current plan or infrastructure in place to support external data requests.